CLINICAL TRIAL: NCT06218017
Title: Development of Algorithm to Precise Monitoring Respiratory Sound During Deep Sedation Using the High Flow Nasal Oxygen System
Brief Title: Development of an Algorithm to Denoise HFNO-generated Tracheal Sound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 202310040DINC
Record Dates: First submitted 2024-01-02; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Endoscopy, Gastrointestinal; Sedation, Conscious
Keywords: Tracheal sound; Electronic auscultation; High flow nasal oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNO first (Experimental): This study follows a crossover design employing a randomized controlled methodology. Patients undergoing gastrointestinal endoscopy and receiving deep sedation were monitored using electronic tracheal sound auscultation. Within this group, patients first underwent a 10-minute session of high-flow nasal oxygen (50 L/min) followed by the utilization of the standard low-flow nasal oxygen (4 L/min). Electronic tracheal sound recordings were obtained during both the high-flow and low-flow nasal oxygen administrations. The aim is to develop an algorithm capable of mitigating the noise generated specifically by the high-flow nasal oxygen.
  Interventions: Device: High flow nasal oxygen fist
- HFNO later (Active Comparator): This study follows a crossover design employing a randomized controlled methodology. Patients undergoing gastrointestinal endoscopy and receiving deep sedation were monitored using electronic tracheal sound auscultation. Within this group, patients first underwent a 10-minute session of standard low-flow nasal oxygen (4 L/min) followed by the utilization of the high-flow nasal oxygen (50 L/min). Electronic tracheal sound recordings were obtained during both the high-flow and low-flow nasal oxygen administrations. The aim is to develop an algorithm capable of mitigating the noise generated specifically by the high-flow nasal oxygen
  Interventions: Device: High flow nasal oxygen later

INTERVENTIONS:
Device: High flow nasal oxygen fist — Patients in the two study group first underwent a 10-minute session of high-flow nasal oxygen (50 L/min) followed by the utilization of the standard low-flow nasal oxygen (4 L/min) or underwent a 10-minute session of standard low-flow nasal oxygen (4 L/min) followed by the utilization of the high-flow nasal oxygen (50 L/min).
  Arms: HFNO first
Device: High flow nasal oxygen later — Patient in this group underwent a 10-minute session of standard low-flow nasal oxygen (4 L/min) followed by the utilization of the high-flow nasal oxygen (50 L/min)
  Arms: HFNO later

SUMMARY:
This study aims to develop an algorithm to mitigate the noise generated by the high-flow nasal oxygen system for tracheal sound monitoring in deeply sedated patients.

DETAILED DESCRIPTION:
During deep sedation without intubation, anesthesia respiratory care and monitoring are of utmost importance. Anesthesia can lead to adverse respiratory effects, increasing the risk of airway obstruction and respiratory depression. High-flow nasal oxygen (HFNO) systems are often used to mitigate these risks. Monitoring tracheal breathing sounds directly using amplification provides better detection accuracy. However, traditional auscultation instruments have limitations, including noise interference and lack of visual functionality. The Airmod Smart Respiratory Monitoring System, with FDA approval in the United States and Taiwan, addresses these issues. It offers respiratory sound recording, noise filtering, event logging, and respiratory rate analysis. Currently, no digital stethoscope on the market can filter out HFNO noise. Therefore, the current study is to develop an algorithm to mitigate the noise generated by the high-flow nasal oxygen system for tracheal sound monitoring in deeply sedated patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective gastroinestinal endoscoy requiring deep sedation

Exclusion Criteria:

* Histories of sleep apnea, chronic obstructive pulmonary disease, or oropharyngeal tumor
* Patient who has a hisotry of previous intraoral surgery, tracheal surgery or pulmonary resection surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Tracheal sound with and without high-flow nasal oxygen will be measured to develop an algorithm to mitigate the high flow nasal oxygen-generated tracheal noise | 20-30 minutes
  We aim to develop an algorithm capable of mitigating the noise generated specifically by the high-flow nasal oxygen based on recording the tracheal sound of patients undergoing gastrointestinal endoscopy in deep sedation with and without high flow nasal oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- National Tawain University Hospital Hsinchu branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared by contacting the principle investigator for rational research purpose.
Supporting Information: Analytic Code
Time Frame: 20-30 min
Access Criteria: By contacting the principle investigator on the basis of rational research purpose.